CLINICAL TRIAL: NCT00376129
Title: Open-Label,Singel Center Study to Evaluate the Safety and Efficacy of an Intramuskcular 12 Week-Course of Alefacept in Patients With Atopic Dermatitis
Brief Title: Open-Label,Singel Center Study of Alefacept in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Biogen-Dompé AG (Industry)
Responsible Party: Prof. Yawalkar, Dermatological Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IST-EU-098-04-AME
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — 15 mg i.m. once weekly for 12 weeks

SUMMARY:
Protocol Title: Open-label,single center study to evaluate the savety and efficacy of an intramuscular 12 week-course of Alefacept in patients with atopic dermatitis.

Study Phase: II

Study Design: Open-label, single center Primary Study Objective: to determine the safety and efficacy of one course of Alefasept when administered as a 15 mg intramuscular ( IM) injektion to patients with atopic dermatitis

Secondary Study Objective: to investigate key immunological parameters involved in the pathology of this common skin disease to interpret the clinical findings

Number of patients: 10

Study Population: Male and female patients, at least 18 years of age with atopic dermatitis, aktive inflammation, a severity score of 6-9 according to Langeland and Rajika and an EASI of >20

Treatment Groups: Alefacept will be administered as a 15 mg IM injection once a week for 12 weeks, followed by a 12-week follow-up period.

DETAILED DESCRIPTION:
Atopic dermatitis is a common chronic eczematous skin disease,wich often begins early in infancy and runs a course of remissions and exacerbations. T-lymphocytes play a prominent role in this skin disease. they represent the majority of skin-infiltrating cells and patients suffering from AD also have increased levels of activated circulating T cells and increased levels of markers of lymphocyte activation such as L-selectin and IL-2R.

ELIGIBILITY:
Inclusion Criteria:

* must give written informed consent
* must be at least 18 years of age
* must have been diagnosed with atopic dermatitis fulfilling the diagnostic criteria of Hanfin und Rajka and having active inflammation
* must have a severity score of 6-9 according to Langeland and Rajka and an EASI of > 20
* must have a PGA of "moderate","severe", or "very severe" and a pruritus score of "moderate" or"severe" at baseline
* must have total lymphocyte counts and CD4+ lymphocyte counts at or above the lower limit of normal

Exclusion Criteria:

* Patients with severe diseases, that might interfere with the evaluation of AD
* Patiens with severe diseases of other organ systems that might put the patient on risk during the study or might interfere with the evaluations
* Patients older than 65 years
* Systemic treatment for atopic dermatitis ( e.g. cyclosporine, mycophenolat- mofetil,inferferon-gamma, PUVA) or systemic treatment with immunosuppressive/immunomodulating substances( e.g. azathioprin,methotrexate,biologics or hyposensitization - therapy) for other indications within 28 days prior to baseline
* local treatment for atopic dermatitis with pimecrolimus/tacrolimus, steroids > class III, unstable use of steroid< class III, emollients or local antiseptics/antibiotics, UVB,UVA within 14 days prior to baseline
* Serious local infection (e.g. cellulitis, abscess)or systemic infection (e.g. pneumonia,septicemia) within 3 months prior to the first dose of Alefacept
* Congenital or acquired immunodeficiency syndrome
* History of an invasive malignancy. Patients with a history of treatmend squamous cell and/or basal call carcinomas limited to the skin are not exluded
* Laboratory or clinical evidence of active tuberculosis
* Current treatment with any therapy for active tuberculosis or tuberculosis prophylaxis
* for female patients, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception, as defined by the investigator, during the study. the rhythm method is not to be used as the sole method of contraception. Female patients considering becoming pregnant while in the study are excluded
* female patients who are currently pregnant or breast-feeding
* abnormal chemistry, i.e., LFTs greater than three times the upper limit of normal
* Current enrollment in any other investigational drug study
* previous participation in this study or previous studies with Alefacept

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
primary endpoints is the change of EASI at Visit 13 compared to baseline via paired t-Test | 24 weeks

SECONDARY OUTCOMES:
Additional enppoints are the percentage of patients reaching a PGA of "clear" or "almost clear" and/or a reduction of EASI of>=50 or >=75% compared to baseline at any visit after baseline. | 24 weeks
the percentage of patients reaching a pruritus score of none or mild | 24 weeks
Several immunological endpoints | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Yawalkar, Prof, Principal Investigator — Dermatological Clinic Berne
Locations (1):
- Inselspital Dermatology, Bern, Canton of Bern, Switzerland